CLINICAL TRIAL: NCT02747719
Title: Effects of Light and Exercise on Human Circadian Rhythms and Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: NSBRI (Unknown)
Responsible Party: Principal Investigator, Elizabeth B. Klerman, Associate Professor, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HFP02802
Record Dates: First submitted 2016-04-18; First posted 2016-04-22 (Estimated); Last update posted 2018-07-11 (Actual); Status verified 2018-07

CONDITIONS: Circadian Rhythm
MeSH Terms: interventions — Light; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Light and exercise (Experimental): Exposure to light with exercise
  Interventions: Behavioral: Light and exercise

INTERVENTIONS:
Behavioral: Light and exercise — Exposure to light and exercise

SUMMARY:
Both light and exercise are effective countermeasures for space and ground-based crews for circadian phase resetting and alertness levels. The investigators propose to test the combined effects of these two countermeasures to determine whether adding exercise to light stimuli will further improve circadian phase resetting and alertness.

ELIGIBILITY:
Inclusion Criteria:

* healthy by history, physical exam, laboratory studies of blood and urine, and psychological screening
* moderate-intensity exercise for at least 150 minutes per week

Exclusion Criteria:

* color blind
* no prescription medications, except hormonal birth control in females

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Circadian Phase | 8 days
  Circadian Phase will be measured using the change in timing of the melatonin rhythm on different days of the protocol. Melatonin will be assayed in blood and/or saliva.

SECONDARY OUTCOMES:
Subjective alertness | 8 days
  Subjective alertness will be measured using the change in values on standardized mood scales on different days of the protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth B Klerman, MD PhD, Principal Investigator — Associate Professor
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided